CLINICAL TRIAL: NCT05563103
Title: Breathing Low Oxygen to Enhance Spinal Stimulation Training and Functional Recovery in Persons With Chronic SCI: The BO2ST Trial
Brief Title: Combination Therapy to Improve SCI Recovery.
Acronym: BO2ST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Randy Trumbower, PT, PhD, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022P002036; W81XWH-22-1-0998 (Other Grant/Funding Number: US Dept. of Defense)
Record Dates: First submitted 2022-09-26; First posted 2022-10-03 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries
Keywords: Walk; Rehabilitation; Strength; Movement; Spinal cord injury; low oxygen; electrical stimulation; walking training
MeSH Terms: conditions — Spinal Cord Injuries | interventions — salicylhydroxamic acid; Walking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AIH + Walking Training with transcutaneous spinal stimulation (WALKtSTIM) (Experimental): Acute Intermittent Hypoxia will be used as a pretreatment before walking training paired with transcutaneous spinal cord stimulation.
  Interventions: Other: Daily acute intermittent hypoxia; Other: Walking + tSTIM
- Sham + WALKtSTIM (Sham Comparator): Sham acute intermittent hypoxia will be used as a pretreatment before walking training paired with transcutaneous spinal cord stimulation.
  Interventions: Other: Room air (SHAM); Other: Walking + tSTIM
- AIH + Walking Training with sham transcutaneous spinal stimulation (WALKtSHAM) (Sham Comparator): Acute Intermittent Hypoxia will be used as a pretreatment before walking training paired with sham transcutaneous spinal cord stimulation.
  Interventions: Other: Daily acute intermittent hypoxia; Other: Walking + Sham transcutaneous spinal stimulation (tSHAM)

INTERVENTIONS:
Other: Daily acute intermittent hypoxia — Each participant will be exposed to 8 sessions of daily acute intermittent hypoxia via air generators over the span of two weeks. The generator will fill reservoir bags attached to a non-rebreathing facemask. Each session will consist of 15 episodes which include intervals of 1.5 minute hypoxia (FIO2=0.10±0.02, i.e. 10% O2) and 1 minute normoxia (FIO2=0.21±0.02).
  Arms: AIH + Walking Training with sham transcutaneous spinal stimulation (WALKtSHAM); AIH + Walking Training with transcutaneous spinal stimulation (WALKtSTIM)
Other: Room air (SHAM) — Each participant will be exposed to 8 sessions of daily room air via air generators over the span of two weeks. The generator will fill reservoir bags attached to a non-rebreathing facemask. Each session will consist of 15 episodes of 1.5 minute normoxia (FIO2=0.21±0.02).
  Arms: Sham + WALKtSTIM
Other: Walking + tSTIM — Individuals will participate in 45 minutes of gait training while having transcutaneous spinal cord stimulation. Stimulation intensity will be 80% involuntary motor threshold.
  Arms: AIH + Walking Training with transcutaneous spinal stimulation (WALKtSTIM); Sham + WALKtSTIM
Other: Walking + Sham transcutaneous spinal stimulation (tSHAM) — Individuals will participate in 45 minutes of gait training while having SHAM transcutaneous spinal cord stimulation. The stimulation will briefly increase to 80% involuntary motor threshold and then brought down to 0 within 30 seconds.
  Arms: AIH + Walking Training with sham transcutaneous spinal stimulation (WALKtSHAM)

SUMMARY:
The purpose of this study is to determine how combining bouts of low oxygen, transcutaneous spinal cord stimulation, and walking training may improve walking function for people with chronic spinal cord injury.

DETAILED DESCRIPTION:
The goal of the study is to determine whether repeatedly breathing mild bouts of low oxygen for brief periods (termed acute intermittent hypoxia (AIH)) combined with transcutaneous spinal cord stimulation (tSTIM) improves recovery of walking and strength after spinal cord injury. This idea stems from animal studies on respiration, in which investigators showed that mild AIH improves breathing in rats with spinal injuries as well as studies involving spinal cord stimulation. These studies showed that AIH induces plasticity, strengthening neural connections by increasing the production of key proteins and improving the sensitivity of spinal cord circuitry. Additional studies have shown that tSTIM may enhance function and strength for people with spinal cord injuries. The ultimate goal of this research is to assess if combining AIH and tSTIM with walking training can enhance individuals walking training greater than just AIH or tSTIM. By using low oxygen as a pre-treatment to tSTIM during walking training, functional independence and quality of life for servicemen and civilians may improve.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age
* medically stable with medical clearance from study physician to participate
* SCI at or below C2 (phrenic sparing) and at or above L2 with at least some sensory or motor function preserved below the neurologic level
* non-progressive etiology of spinal injury
* American Spinal Injury Association (ASIA) scores of C-D at initial screen
* ambulatory (able to complete the 10-meter walk test without support from another person)
* chronic injury (define as > 12 months post-injury) to avoid potential for spontaneous neurological plasticity and recovery

Exclusion Criteria:

* severe concurrent illness or pain, including unhealed decubiti, severe neuropathic or chronic pain syndrome, severe infection (e.g., urinary tract), hypertension, cardiovascular disease, pulmonary disease, severe osteoporosis, active heterotopic ossification in the lower extremities, severe systemic inflammation
* < 24 on Mini-Mental Exam
* severe recurrent autonomic dysreflexia
* history of severe cardiovascular/pulmonary complications including hypertension (systolic blood pressure > 150 mmHg)
* pregnancy because of unknown effects of AIH or tSTIM on a fetus (individuals of childbearing potential will not otherwise be excluded)
* botulinum toxin injections in lower extremity muscles within the prior three months
* history of tendon or nerve transfer surgery in the lower extremity
* untreated severe sleep-disordered breathing characterized by uncontrolled hypoxia and sleep fractionation that may impact the outcome of this study.
* active implanted devices (e.g., intrathecal baclofen pump)
* receiving concurrent electrical stimulation
* motor threshold evoked by transcutaneous spinal stimulation >200 mA

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in walking recovery, assessed by 10 meter walk test (10MWT) | Through study completion, an average of 12 weeks
  Participants walk ten meters without assistance at their fastest, but safest speed with a minimum of 1-minute of rest between two trials. Average speed across the up to three 10MWT trials will be used for analysis. Change is the difference between the post-treatment assessment 2 and pre-treatment baseline.
Rate of change in walking recovery, assessed by 10 meter walk test (10MWT) | Through study completion, an average of 12 weeks
  Participants walk ten meters without assistance at their fastest, but safest speed with a minimum of 1-minute of rest between two trials. Average speed across the up to three 10MWT trials will be used for analysis. Rate of change is the number of treatment sessions required to achieve an increase in 10MWT speed of at least the minimal clinically important difference (0.06 m/s) as compared to pre-treatment baseline.

SECONDARY OUTCOMES:
Change in walking recovery, assessed by 6 minute walk test (6MWT) | Through study completion, an average of 12 weeks
  Participants perform the 6MWT at their fastest, most comfortable walking speed sustainable for 6 minutes. Distances will be recorded at 2 and 6 minutes. The test will be based upon the participant's ability to finish each assessment without human assistance. Change is the difference between the post-treatment assessment 2 and pre-treatment baseline.
Change in walking recovery, assessed by timed up-and-go (TUG) test | Through study completion, an average of 12 weeks
  The TUG test is used to assess the dynamic balance of an individual. It measures the amount of time (recorded in seconds) it takes for the individual to rise from a standard arm chair, walk a distance of 3 meters and return to the initial position resting against the back of the chair. Participants will perform up to three trials of the TUG test. Average speed across TUG trials will be used for analysis. Change is the difference between the post-treatment assessment 2 and pre-treatment baseline.
Change in pain severity, assessed by the Numeric Pain Rating Scale (NPRS) | Through study completion, an average of 12 weeks
  Participants will report their pain level using the Numeric Pain Rating Scale. The scale is from 0 to 10; 0 being no pain and 10 being extreme pain. Change is the difference between the post-treatment assessment 2 and pre-treatment baseline.
Change in cognitive function, assessed by the California Verbal Learning Test (CVLT) | Through treatment completion, an average of 4 weeks
  The CVLT is a brief, individually administered battery to measure cognitive decline or improvement and assesses verbal learning and memory for older adolescents and adults. Change is the difference between the post-treatment assessment 2 and pre-treatment baseline.
Systemic hypertension incidence rate | Through treatment completion, an average of 4 weeks
  Participants will have their systolic and diastolic blood pressure measured. A systemic hypertensive event is quantified as a systolic pressure exceeding 140 mmHg and/or diastolic pressure exceeding 90 mmHg. A hypertension incident rate is the number of hypertensive events divided by the total person-time. Person-time is in units of person-measures (the sum of the total number of BP measurements) taken for each person. Person-measures accounts for the total number of chances for detecting a hypertensive event and accounts for measurements not made due to drop-out or a disqualifying adverse event.
Autonomic dysreflexia incidence rate | Through treatment completion, an average of 4 weeks
  The occurrence of autonomic dysreflexia will be assessed. An autonomic dysreflexia event will constitute a participant having a SBP increase from baseline of 20 mmHg not associated with exercise or systolic blood pressure (SBP) greater than 150 mmHg with complaints of headache, diaphoresis, and/or blurred vision and will be diagnosed by our study team clinicians. We will compute autonomic dysreflexia incident rate as the number of autonomic dysreflexia events divided by the total person-time. We define person-time in units of person-days (the number of days a person remains in the study). Person-days account for the total number of chances for detecting autonomic dysreflexia and accounts for days on which measurements were not made due to drop-out or a disqualifying adverse event.

OTHER OUTCOMES:
Change in lower extremity strength, assessed by American Spinal Injury Association Impairment Scale (AIS) lower extremity motor scores (LEMS) | Through study completion, an average of 12 weeks
  The LEMS uses ASIA key muscles in both the lower extremities, with a total possible score of 50 (maximum score of 5 for each muscle group). Change is the difference between the post-treatment assessment 2 and pre-treatment baseline.
Change in spasticity, assessed by the Spinal Cord Assessment Tool for Spastic Reflexes (SCATS) | Through study completion, an average of 12 weeks
  The study team will quantify the total lower extremity spasticity score using the cumulative sum of 3 SCATS subscales: clonus (0=no spasticity; 3=severe), flexor (0=no spasticity; 3=severe), and extensor (0=no spasticity; 3=severe). Change is the difference between the post-treatment assessment 2 and pre-treatment baseline.
Change in bowel dysfunction, assessed by the Neurogenic Bowel Dysfunction Score (NBDS) v2.1 | Through study completion, an average of 12 weeks
  This questionnaire is a symptom-based score for neurogenic bowel dysfunction. Change is the difference between the post-treatment assessment 2 and pre-treatment baseline.
Change in bladder dysfunction, assessed by the Neurogenic Bladder Symptom Score (NBSS) | Through study completion, an average of 12 weeks
  This questionnaire is a symptom-based score for neurogenic bladder dysfunction. Change is the difference between the post-treatment assessment 2 and pre-treatment baseline.
Change in walking ability and assistive device use, assessed by Spinal Cord Injury Functional Ambulation Inventory (SCI-FAI). | Through study completion, an average of 12 weeks
  The SCI-FAI assesses functional walking ability in ambulatory individuals with SCI. Component scores range from 0 to 20 in the gait parameter component, 0 to 14 in the assistive device component, and 0 to 5 in the walking mobility component. Change is the difference between the post-treatment assessment 2 and pre-treatment baseline.
Change in physical assistance needed, assessed by Walking Index for Spinal Cord Injury (WISCI) II | Through study completion, an average of 12 weeks
  The WISCI is used to assess the amount of physical assistance is needed as well as devices required for walking following paralysis. This assessment is from 0-20 with value corresponding to a physical assistance description. Change is the difference between the post-treatment assessment 2 and pre-treatment baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Randy Trumbower, PT, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (2):
- United States (2):
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - Spaulding Rehabilitation Hospital, Cambridge, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be available to other researchers upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol and statistical analysis plan will be disseminated by December 2022. Participant data will be available at the end of the trial.
Access Criteria: Principal investigators will be able to receive deidentified data.

REFERENCES:
- [Background] Cutler MJ, Swift NM, Keller DM, Wasmund WL, Smith ML. Hypoxia-mediated prolonged elevation of sympathetic nerve activity after periods of intermittent hypoxic apnea. J Appl Physiol (1985). 2004 Feb;96(2):754-61. doi: 10.1152/japplphysiol.00506.2003. Epub 2003 Oct 10. PMID 14555683
- [Background] Dale-Nagle EA, Hoffman MS, MacFarlane PM, Mitchell GS. Multiple pathways to long-lasting phrenic motor facilitation. Adv Exp Med Biol. 2010;669:225-30. doi: 10.1007/978-1-4419-5692-7_45. PMID 20217354
- [Background] Estes S, Zarkou A, Hope JM, Suri C, Field-Fote EC. Combined Transcutaneous Spinal Stimulation and Locomotor Training to Improve Walking Function and Reduce Spasticity in Subacute Spinal Cord Injury: A Randomized Study of Clinical Feasibility and Efficacy. J Clin Med. 2021 Mar 11;10(6):1167. doi: 10.3390/jcm10061167. PMID 33799508
- [Background] Gad P, Hastings S, Zhong H, Seth G, Kandhari S, Edgerton VR. Transcutaneous Spinal Neuromodulation Reorganizes Neural Networks in Patients with Cerebral Palsy. Neurotherapeutics. 2021 Jul;18(3):1953-1962. doi: 10.1007/s13311-021-01087-6. Epub 2021 Jul 9. PMID 34244928
- [Background] Tan AQ, Sohn WJ, Naidu A, Trumbower RD. Daily acute intermittent hypoxia combined with walking practice enhances walking performance but not intralimb motor coordination in persons with chronic incomplete spinal cord injury. Exp Neurol. 2021 Jun;340:113669. doi: 10.1016/j.expneurol.2021.113669. Epub 2021 Feb 27. PMID 33647273
- [Background] Hayes HB, Jayaraman A, Herrmann M, Mitchell GS, Rymer WZ, Trumbower RD. Daily intermittent hypoxia enhances walking after chronic spinal cord injury: a randomized trial. Neurology. 2014 Jan 14;82(2):104-13. doi: 10.1212/01.WNL.0000437416.34298.43. Epub 2013 Nov 27. PMID 24285617
- [Background] Trumbower RD, Jayaraman A, Mitchell GS, Rymer WZ. Exposure to acute intermittent hypoxia augments somatic motor function in humans with incomplete spinal cord injury. Neurorehabil Neural Repair. 2012 Feb;26(2):163-72. doi: 10.1177/1545968311412055. Epub 2011 Aug 5. PMID 21821826
- [Derived] Muter WM, Mansson L, Tuthill C, Aalla S, Barth S, Evans E, McKenzie K, Prokup S, Yang C, Sandhu M, Rymer WZ, Edgerton VR, Gad P, Mitchell GS, Wu SS, Shan G, Jayaraman A, Trumbower RD. A Research Protocol to Study the Priming Effects of Breathing Low Oxygen on Enhancing Training-Related Gains in Walking Function for Persons With Spinal Cord Injury: The BO2ST Trial. Neurotrauma Rep. 2023 Nov 6;4(1):736-750. doi: 10.1089/neur.2023.0036. eCollection 2023. PMID 38028272